CLINICAL TRIAL: NCT06814574
Title: Pacemaker Implantation Following Transcatheter Tricuspid Valve Replacement - Single Center Experience
Brief Title: Pacemaker Implantation Following Transcatheter Tricuspid Valve Replacement
Status: Recruiting | Type: Observational
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Other Study IDs: GER-EP-26
Record Dates: First submitted 2025-01-28; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: AV Block Complete; Tricuspid Regurgitation (TR)
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
Transcatheter tricuspid valve replacement (TTVR) is associated with a high risk of third-degree atrioventricular block (AVB). However, the optimal pacemaker management following TTVR remains unclear. This study aims to identify an optimal therapeutic approach for pacemaker implantation in patients undergoing TTVR.

ELIGIBILITY:
Inclusion Criteria:

* Transcatheter Tricuspid Valve Replacement

Exclusion Criteria:

* no defined exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include every patient with a transcatheter tricuspid valve replacement in the study period.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Success | at the time of surgery
  The number of patients in whom the initially chosen pacemaker implantation approach was successfully performed, relative to all pacemaker implantations following TTVI.
Feasibility | at the time of surgery
  Successful pacemaker implantation, regardless of the type of pacemaker, in relation to all patients with a relevant indication following TTVR.
Safety | through study completion (an average of 6 Months)
  Peri- and postprocedural complications associated with pacemaker implantation after TTVR.

SECONDARY OUTCOMES:
Type of Pacemaker Implantation | at the time of surgery
  eg. Leadless, right ventricular lead, coronary sinus lead, epicardial lead
Pacemaker Implantation - Procedural Details | at the time of surgery
  Procedural Details of the pacemaker Implantation, e.g. Fluoroscopy Time, OP-Duration.
Electric Performance | at the time of surgery, through study completion (an average of 6 Months)
  Performance of the electrical pacemaker parameters (e.g. Sensing, Stimulation Threshold, Impedance). Intraoperative measurements and routine device-interrogations in follow-Up.

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzentrum München, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes